CLINICAL TRIAL: NCT01166451
Title: Iron Deficiency Anemia and Infant Behavior: Preventive Trial
Brief Title: The Anemia Control Program: High or Low Iron Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Betsy Lozoff, MD, Professor of Pediatrics and Communicable Diseases and Research Professor, Center for Human Growth and Development, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01HD033487 (NIH)
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Iron Deficiency Anemia; Cognitive Development; Motor Development
Keywords: iron deficiency anemia; cognitive development; motor development
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Low-iron (Experimental): Infants randomly assigned at 6 months of age to receive low-iron formula (average 2.3 mg/L, range 1.6 - 2.4 mg/L) until 12 months of age.
  Interventions: Dietary Supplement: Low-iron formula
- High-iron (Experimental): Infants randomly assigned at 6 months of age to receive high-iron formula (average 12.7 mg/L) until 12 months of age.
  Interventions: Dietary Supplement: High-iron formula

INTERVENTIONS:
Dietary Supplement: Low-iron formula — Infants randomly assigned at 6 months of age to receive low-iron formula (average 2.3 mg/L, range 1.6 - 2.4 mg/L) until 12 months of age. Low-iron formula distributed in powdered form. Project personnel visited infants' homes weekly to record measures of powdered formula used per day. Formula consumption was also verified by the number of cans given by the clinic nurse at each visit (regular pediatric visits and monthly clinic appointments until 12 months of age.)
  Arms: Low-iron
Dietary Supplement: High-iron formula — Infants randomly assigned at 6 months of age to receive high-iron formula (average 12.7 mg/L) until 12 months of age. High-iron formula distributed in powdered form. Project personnel visited infants' homes weekly to record measures of powdered formula used per day. Formula consumption was also verified by the number of cans given by the clinic nurse at each visit (regular pediatric visits and monthly clinic appointments until 12 months of age.)
  Arms: High-iron

SUMMARY:
The purpose of this clinical trial was to determine if high-iron or low-iron formula, containing an average of 12.7 mg/L or 2.3 mg/L respectively, had differing effects on iron status in infancy and on development longitudinally.

DETAILED DESCRIPTION:
For a detailed description of the clinical trial setting and procedures in infancy, please refer to the following:

Walter T, Pino P, Pizarro F and Lozoff B. Prevention of iron-deficiency anemia: Comparison of high- and low-iron formulas in term healthy infants after six months of life. J Pedr 1998:132:635-40.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight >= 3.0 kg
* single birth
* no major congenital anomalies
* no major birth or neonatal complications
* no emergency c-section
* no jaundice requiring phototherapy
* no hospitalization for more than 5 days
* no chronic illness
* no iron therapy
* already started to received some bottle feedings by 6 months of age

Exclusion Criteria:

* residence outside identified neighborhoods
* another infant <12 months in household
* infant in daycare
* unstable, illiterate, or psychotic caregiver

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 835 (Actual)
Dates: Start 1991-09; Primary Completion 1994-08 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Iron deficiency anemia | 12 and 18 months

SECONDARY OUTCOMES:
Longitudinal child behavior and development | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Lozoff, MD, Principal Investigator — University of Michigan
Locations (1):
- Instituto de Nutriticion y Tecnologia de los Alimentos, Santiago, Chile

REFERENCES:
- [Result] Walter T, Pino P, Pizarro F, Lozoff B. Prevention of iron-deficiency anemia: comparison of high- and low-iron formulas in term healthy infants after six months of life. J Pediatr. 1998 Apr;132(4):635-40. doi: 10.1016/s0022-3476(98)70352-x. PMID 9580762
- [Derived] East PL, Reid B, Blanco E, Burrows R, Lozoff B, Gahagan S. Iron supplementation given to nonanemic infants: neurocognitive functioning at 16 years. Nutr Neurosci. 2023 Jan;26(1):40-49. doi: 10.1080/1028415X.2021.2013399. Epub 2021 Dec 19. PMID 34927561
- [Derived] East P, Doom J, Blanco E, Burrows R, Lozoff B, Gahagan S. Young adult outcomes associated with lower cognitive functioning in childhood related to iron-fortified formula in infancy. Nutr Neurosci. 2022 Apr;25(4):709-718. doi: 10.1080/1028415X.2020.1804099. Epub 2020 Aug 11. PMID 32778008
- [Derived] Gahagan S, Delker E, Blanco E, Burrows R, Lozoff B. Randomized Controlled Trial of Iron-Fortified versus Low-Iron Infant Formula: Developmental Outcomes at 16 Years. J Pediatr. 2019 Sep;212:124-130.e1. doi: 10.1016/j.jpeds.2019.05.030. Epub 2019 Jun 26. PMID 31253407
- [Derived] Lozoff B, Castillo M, Clark KM, Smith JB. Iron-fortified vs low-iron infant formula: developmental outcome at 10 years. Arch Pediatr Adolesc Med. 2012 Mar;166(3):208-15. doi: 10.1001/archpediatrics.2011.197. Epub 2011 Nov 7. PMID 22064877